CLINICAL TRIAL: NCT01377402
Title: ARgentinean Risk Assessment Registry in Acute Coronary Syndrome; the ARRA-RACS Study.
Brief Title: ARgentinean Risk Assessment Registry in ACS; the ARRA-RACS Study
Acronym: ARRA-RACS
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Universidad Católica de Salta (Unknown)
Responsible Party: Sponsor
Other Study IDs: ARRA-RACS
Record Dates: First submitted 2011-06-20; First posted 2011-06-21 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Chest Pain; Coronary Artery Disease; Unstable Angina Pectoris; Myocardial Infarction
MeSH Terms: conditions — Chest Pain; Coronary Artery Disease; Angina, Unstable; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Citrated plasma, EDTA-plasma and packed red blood cells are kept in suitable aliquots at -80 degrees Celcius.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chest pain: Men and women admitted with chest pain and suspected acute coronary syndrome (ACS).

SUMMARY:
The first aim of this trial is to assess the long-term prognostic value of Omega-3 index, which is a measure of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) relative to other fatty acids in the erythrocyte membrane, in an unselected, regional multicenter observational study of 982 chest pain patients admitted to the emergency unit, employing blood samples collected at admission.

The second purpose of this study is to evaluate the prognostic utility of vitamin D in the same population.

The third purpose of this study is to assess the incremental prognostic value of B-type natriuretic peptide (BNP) and high-sensitive C-reactive protein (hsCRP).

DETAILED DESCRIPTION:
BACKGROUND Cardiac troponins are sensitive markers for myocardial injury in ACS and even a minor elevation of cardiac troponins is associated with an increased risk for future adverse coronary events. However, a detectable troponin release occurs only in a part of patients admitted with ACS. The clinical outcomes and further prognosis of patients with ACS with absent TnT release vary widely, and the identification of potential high-risk patients with troponin negative ACS still remains a major problem in clinical routine. Therefore, the aim of this study is focused on identifying new biomarkers for risk stratification.

Omega- 3 Index: The value of the Omega-3 Index as a prognostic marker in the acute coronary syndromes is still under investigation.

Vitamin D deficiency is positively correlated with cardiovascular risk and N-3 polyunsaturated fatty acids (PUFA's) may reduce the risk of cardiovascular disease. Vitamin D can either be ingested, or created in the skin on exposure to sun, whereas PUFA's are largely incorporated through the diet. Vitamin D deficiency in humans is increasing and its levels are influenced by the color of the skin, geographical location, latitude, altitude, season and daytime.

In addition to Vitamin D, several studies have shown that, N-3 polyunsaturated fatty acids (PUFA's), also have a positive impact on the cardiovascular system. PUFA's are not sufficiently synthesized in the body and are incorporated through the diet. These essential fatty acids are found almost exclusively in oily fish, and have been shown to have a positive impact on several cardiovascular risk factors.

Fish, a source of both Vitamin D and omega-3, is frequently consumed by the costal population of Norway, and is less preferred by the inland beef-consuming population in Northern Argentina. The subtropical location and altitude of Salta, Argentina, is associated with a higher exposure to sun in comparison to the temperate location of Norway. The uptake of Vitamin D in the costal population of Norway may essentially be through the diet, whereas sun exposure may be the essential source of Vitamin D in the Northern Argentinean population.

By investigating the correlation between omega-3 and Vitamin D, we may better understand the nutritional impact on Vitamin D and its correlation with n-3 PUFA's.

B-type natriuretic peptide: B-type natriuretic peptide (BNP) is a counter-regulatory peptide hormone predominantly synthesized in the ventricular myocardium. BNP is released into the circulation in response to ventricular dilatation and pressure overload, and reflects ventricular wall stress and tissue hypoxia rather than cell injury per se. It is a well known marker of left ventricular dysfunction and heart failure (HF), and it provides prognostic information beyond and above left ventricular ejection fraction (LVEF) in patients with an acute coronary syndrome (ACS). This marker of neurohormonal activation and inflammation plays a pivotal role across the spectrum of ACS, including patients with ST-elevation myocardial infarction (MI) and non ST-elevation ACS (NSTE-ACS). Previous studies have demonstrated that BNP measured in the first days after the onset of symptoms independently predicts mortality, HF, and new MI in this patient population. Elevated natriuretic peptides at presentation have been shown to identify patients with ACS who are at higher risk of death and HF, and it adds information to that provided by the troponins. However, in a low-risk population the association between elevated BNP and survival is attenuated when adjustment is made for echocardiographic variables (in addition to clinical covariates), as shown by Wang and colleagues. In addition, they did not find any association between baseline BNP and the risk of coronary heart disease (CHD).

High-sensitive C-reactive protein (hsCRP): C-reactive protein (CRP) is an acute-phase reactant that is produced in response to acute injury, infection or other inflammation stimuli. It is a marker for underlying systemic inflammation and plays an important role in the initiation and propagation of atherosclerosis and ultimately to plaque rupture and the ensuing thrombotic complication. Elevated levels of CRP were first reported in patients hospitalized with NSTE-ACS in the early 1990s. Through the use of appropriate high-sensitive assays, it has been possible to investigate the relationship between plasma CRP levels that previously were considered to be normal and cardiovascular disease (CVD). Nevertheless, it is still under debate which markers should be preferred for risk prediction. It has been suggested that the combined evaluation of BNP and CRP may yield incremental prognostic information in the risk stratification of patients with ACS, and their combined use has been shown to improve long-term risk prediction of mortality in patients with stable CHD. To our knowledge, there are limited data available that directly compare these two markers in a prospective manner in an unselected patient population presenting to the emergency department (ED) with chest pain. In addition, their role in risk stratification in patients with ACS is still under evaluation, and therefore additional investigations are necessary.

STUDY DESIGN This prospective regional multicenter observational non-invasive trial includes 982 men and women admitted with chest pain and potential ACS at nine hopitals in Salta, Argentina between November 2005 and November 2008. Blood samples were collected immediately following admission. Patients were stratified according to peak troponin T (TnT) release following admission; i.e. 1) patients with an admission TnT exceeding 0.01 ng/mL, and 2) patients with a TnT level below 0.01 ng/mL.

Assessment of a history of previous MI, angina pectoris (AP), congestive heart failure (CHF), diabetes mellitus and arterial hypertension was based on hospital records and personal interview. Electrocardiographic findings at admission were classified according to the presence of ST segment changes.

Written informed consent was obtained from all patients. Survival status, date and cause of death and clinical data were obtained by telephone interview and hospital journal reports at 4 predefined time points (30 days, 6, 12 and 24 months) during the two year follow-up period. In case of incapacity to provide information, the general practitioner or nursery home were contacted for relevant data. Hospital journals were searched for confirmation of reported data.

DATA OWNERSHIP AND PUBLICATION OF RESULTS. The ARRA-RACS Steering Committee has the ownership of all data registered in the ARRA-RACS database, and any use of these data including the preparation and publication of scientific reports must be approved by the Steering Committee. Scientific articles will be published by ARRA-RACS investigators or by authors mentioned by name. The author sequence should be approved by the Steering Committee and based upon contribution. Incentives to involve articles as part of a doctoral thesis should be encouraged. All collaborators in the study will be mentioned by name in an Appendix section of the main article from the study. The results will be published in peer-reviewed scientific journals and in magazines for the general public.

ELIGIBILITY:
Inclusion Criteria:

* adults > 18 years able to give informed consent
* a history of chest pain or other symptoms suggestive of an ACS leading to admission at the emergency unit

Exclusion Criteria:

* < 18 years of age
* Unwillingness or incapacity to provide informed consent
* Prior admission resulting in inclusion in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 982 men and women admitted with chest pain and potential acute cornary syndrome (ACS) at nine hopitals in Salta, Argenitna between November 2005 and November 2008.
Sampling Method: Probability Sample
Enrollment: 982 (Actual)
Dates: Start 2005-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis WT Nilsen, MD PhD Prof., Principal Investigator — Helse Stavanger HF
Locations (10):
- Argentina (9):
  - Clinica Güemes, Salta, Salta Province
  - Clinica San Rafael, Salta, Salta Province
  - Hospital Militar Salta, Salta, Salta Province
  - Hospital Privado Santa Clara de Asis, Salta, Salta Province
  - Hospital San Bernardo, Salta, Salta Province
  - Intituto CENESA, Salta, Salta Province
  - Sanatorio El Carmen, Salta, Salta Province
  - Sanatorio El Parque, Salta, Salta Province
  - Sanatorio San Roque, Salta, Salta Province
- Stavanger University Hospital, Stavanger, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leon de la Fuente R, Naesgaard PA, Nilsen ST, Woie L, Aarsland T, Gallo P, Grundt H, Staines H, Nilsen DW. B-type natriuretic peptide and high sensitive C-reactive protein predict 2-year all cause mortality in chest pain patients: a prospective observational study from Salta, Argentina. BMC Cardiovasc Disord. 2011 Sep 29;11:57. doi: 10.1186/1471-2261-11-57. PMID 21958326
- [Result] de la Fuente RL, Naesgaard PA, Nilsen ST, Woie L, Aarsland T, Gundersen T, Nilsen DW. Omega-3 index and prognosis in acute coronary chest pain patients with a low dietary intake of omega-3. Scand Cardiovasc J. 2013 Apr;47(2):69-79. doi: 10.3109/14017431.2012.747220. Epub 2012 Dec 12. PMID 23127172
- [Result] Leon de la Fuente RA, Naesgaard PA, Nilsen ST, Woie L, Aarsland T, Staines H, Nilsen DW. Socioeconomic assessment and impact of social security on outcome in patients admitted with suspected coronary chest pain in the city of salta, Argentina. Cardiol Res Pract. 2013;2013:807249. doi: 10.1155/2013/807249. Epub 2013 May 29. PMID 23819097
- [Result] Naesgaard PA, Leon de la Fuente RA, Nilsen ST, Woie L, Aarsland T, Staines H, Nilsen DW. Vitamin d predicts all-cause and cardiac mortality in females with suspected acute coronary syndrome: a comparison with brain natriuretic Peptide and high-sensitivity C-reactive protein. Cardiol Res Pract. 2013;2013:398034. doi: 10.1155/2013/398034. Epub 2013 Nov 17. PMID 24349821
- [Result] Nilsen DW, Mjelva OR, Leon de la Fuente RA, Naesgaard P, Ponitz V, Brugger-Andersen T, Grundt H, Staines H, Nilsen ST. Borderline Values of Troponin-T and High Sensitivity C-Reactive Protein Did Not Predict 2-Year Mortality in TnT Positive Chest-Pain Patients, Whereas Brain Natriuretic Peptide Did. Front Cardiovasc Med. 2015 Apr 8;2:16. doi: 10.3389/fcvm.2015.00016. eCollection 2015. PMID 26664888
- [Derived] Aarsetoy R, Ueland T, Aukrust P, Michelsen AE, Leon de la Fuente R, Grundt H, Staines H, Nygaard O, Nilsen DWT. Complement component 7 is associated with total- and cardiac death in chest-pain patients with suspected acute coronary syndrome. BMC Cardiovasc Disord. 2021 Oct 14;21(1):496. doi: 10.1186/s12872-021-02306-w. PMID 34649504
- [Derived] Aarsetoy R, Ueland T, Aukrust P, Michelsen AE, de la Fuente RL, Ponitz V, Brugger-Andersen T, Grundt H, Staines H, Nilsen DWT. Angiopoietin-2 and angiopoietin-like 4 protein provide prognostic information in patients with suspected acute coronary syndrome. J Intern Med. 2021 Oct;290(4):894-909. doi: 10.1111/joim.13339. Epub 2021 Jul 8. PMID 34237166
- [Derived] Naesgaard PA, Leon De La Fuente RA, Nilsen ST, Woie L, Aarsland T, Brede C, Staines H, Nilsen DW. Serum 25(OH)D is a 2-year predictor of all-cause mortality, cardiac death and sudden cardiac death in chest pain patients from Northern Argentina. PLoS One. 2012;7(9):e43228. doi: 10.1371/journal.pone.0043228. Epub 2012 Sep 6. PMID 22970121

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Suspected Acute Coronary Chest Pain: Men and women admitted with chest pain and suspected acute coronary syndrome (ACS).
Period: Overall Study
Arm/Group | Patients With Suspected Acute Coronary Chest Pain
Started | 982
Completed | 982
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with suspected ACS.
Groups:
- Patients With Suspected Acute Coronary Chest Pain: Patients recruited immediately following acute hospital admission for suspected coronary chest pain.
Arm/Group | Patients With Suspected Acute Coronary Chest Pain
Number analyzed (Participants) | 982
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 544
  >=65 years | 438
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [53 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 394
  Male | 588
Region of Enrollment [Number; unit: participants]
  Argentina | 982

OUTCOME MEASURES:

1. Primary Outcome: Total Mortality.
Description: Mortality for any reason
Time Frame: 2-5 years
Population: Patients with suspected ACS
Measure: Number; unit: participants
Groups:
- Patients With Suspected ACS: Patients with acute hospitalisation due to suspected coronary chest pain.
Arm/Group | Patients With Suspected ACS
Number analyzed (Participants) | 982
participants | 173

2. Secondary Outcome: Participants With Cardiac Events During Follow-up.
Description: Cardiovascular Death. Myocardial infarctions (re-MIs) defined according to WHO criteria of 1979.
Time Frame: 2-5 years
Measure: Number; unit: Participants
Groups:
- Cardiovascular Death: Patients with confirmed cardiovascular death during the course of the study
- Myocardial Re-infarction: Patients with one or more myocardial re-infarctions during the course of the study
Arm/Group | Cardiovascular Death | Myocardial Re-infarction
Number analyzed (Participants) | 982 | 982
Participants | 92 | 51

ADVERSE EVENTS:
Description: The study subjects were interviewed at pre-dedetermined intervals from inclusion until end of follow-up.
Groups:
- Patients With Suspected ACS: Patients admitted to hospital with acute chest pain.
Arm/Group | Patients With Suspected ACS
Serious Adverse Events (participants affected / at risk) | 0/982
Other Adverse Events (participants affected / at risk) | 0/982

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes